CLINICAL TRIAL: NCT03195192
Title: Utilizing Multiomic Advanced Diagnostics to Identify CDK 4/6 Inhibitor Response Predictors and a Post-treatment Multiomic Signature for Patients With ER+/HER2- Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Side-Out Foundation (Other)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SO-BCA-003
Record Dates: First submitted 2017-06-09; First posted 2017-06-22 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): This is a biomarker study analyzing tissue for baseline biomarkers and collecting tissue at progression for further analysis of biomarkers changes after treatment with CDK 4/6 inhibitors and endocrine therapy
  Interventions: Other: biomarker study

INTERVENTIONS:
Other: biomarker study — This is a biomarker study

SUMMARY:
This is an open-label, multicenter study in patients with metastatic breast cancer who are candidates for standard first line treatment with palbociclib or ribociclib plus endocrine therapy. To be eligible, patients must have received no prior chemotherapeutic or hormonal regimen for metastatic disease. However, patients may still be considered eligible if they have already started treatment with endocrine therapy (an aromatase inhibitor or fulvestrant) plus palbociclib or ribociclib for no longer than 4 weeks prior to study enrollment, as long as they meet all other eligibility criteria. Eligible patients must have had a diagnostic biopsy of the metastatic lesion no more than 4 months prior to study enrollment and with sufficient tissue to complete the proposed biomarker analysis. Patients who develop disease progression within the first 12 months of starting palbociclib or ribociclib plus endocrine therapy will be eligible for an optional additional tissue biopsy at time of disease progression to repeat the analysis at time of disease progression and obtain real-time (10-14-day turn-around) multi-omic data produced under College of American Pathologist (CAP)/Clinical Laboratory Improvement Amendments (CLIA) development and/or compliant practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease.
* Tumors must be estrogen and/or progesterone receptor positive according to ASCO/CAP 2010 guidelines as either ER or PR ≥ 1% positive nuclear staining by immunohistochemistry based on local laboratory results.
* Tumors must be HER2 negative as defined according to ASCO/CAP 2013, as HER2 0 - 1+ by IHC or non-amplified FISH or CISH. If HER2 IHC is 2+, FISH/CISH must be performed and must not be positive (HER2/CEP17 ratio must be < 2, and HER2 copy number < 6 signals/cell), but otherwise FISH/CISH is not required if IHC is 0 or 1+ by institutional standards.
* Must be candidates to receive endocrine therapy and palbociclib or ribociclib as first-line treatment for their advanced disease. Patients will be considered eligible for study enrollment if they have started on treatment with a standard dose and schedule of palbociclib or ribociclib and endocrine therapy (aromatase inhibitor or fulvestrant) as long as they have not started palbociclib or ribociclib treatment for longer than 4 weeks from time of study enrollment, have sufficient tissue to perform the proposed tissue analysis and must meet all other eligibility criteria. Endocrine therapy can be initiated up to 4 weeks prior to starting palbociclib or ribociclib.
* Patients must have measurable disease by RECIST v.1.1 or bone disease as their only site of disease (with bone lesions confirmed by CT, MRI or bone X-ray).
* No prior treatment with chemotherapy for a diagnosis of locoregionally recurrent or metastatic breast cancer is allowed.
* Be ≥ 18 years of age
* Have an ECOG score of 0-1
* Postmenopausal women defined as women with:

  * Prior bilateral surgical oophorectomy, or
  * Medically confirmed post-menopausal status defined as spontaneous cessation of regular menses for at least 12 consecutive months or follicle-stimulating hormone (FSH), luteinizing hormone (LH) and estradiol blood levels in their respective postmenopausal ranges.
* Premenopausal women will be considered eligible for study participation if they are receiving medical ovarian suppression with luteinizing hormone-releasing hormone (LHRH) agonists with documented estradiol blood levels in their respective postmenopausal ranges.
* Archive tumor tissue (obtained from a biopsy or surgical resection of a metastatic lesion done within 4 months from study enrollment) availability is required for patient participation. If the available tissue is insufficient for the required baseline analysis, the patients are given the option to repeat the biopsy for the purpose of study participation as long as they have not already started palbociclib or ribociclib.
* Understand and provide written informed consent prior to initiation of any study-specific procedures.

Exclusion Criteria:

* Lack of archive tumor tissue from a biopsy or surgical resection of a metastatic lesion done within 4 months of study enrollment. Patients will be given an option to have a repeated biopsy of a metastatic lesion if they had a diagnostic tumor biopsy intended for use in the current study that was performed more than 4 months prior to analysis, or there is insufficient tissue from the initial biopsy to complete the analysis, as long as they have not started treatment with a CDK 4/6 inhibitor. Otherwise, the patient will be excluded from the study participation.
* Have symptomatic CNS metastasis. Patients with a history of CNS metastases who have been treated with whole brain irradiation must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable does of steroids for ≥ 4 weeks prior to enrollment.
* Have uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or ability to willingly give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate baseline phosphorylated RB levels in tumor tissue as a predictive marker of response to palbociclib or ribociclib as first line treatment for ER+/HER2- metastatic breast cancer | 2 years
  Establish baseline values in tumor tissue to use as predictive markers

SECONDARY OUTCOMES:
Evaluate baseline biomarkers which are direct substrates of CDK 4/6 or controlled secondarily by CDK 4/6 kinase activity as qualifying predictive markers of response to CDK 4/6 inhibitors as first line treatment for ER+/HER2- metastatic breast cancer | 2 years
  Identify CDK 4/6 kinase which are either direct substrates or controlled secondarily by CDK 4/6 activity.
Evaluate tumor tissue collected at time of disease progression, for post CDK 4/6 inhibitor treatment changes in biomarkers which are either direct substrates of Cyclin Dependent (CDK) 4/6 kinase or controlled secondarily by CDK 4/6 kinase activity. | 2 years
  Evaluate tissue collected at progression for changes in CDK 4/6 biomarkers after treatment with CDK 4/6 inhibitors.
Evaluate tumor tissue collected at time of disease progression for measurement of the activation state signaling pathways that are known markers for endocrine resistance (e.g. AKT-mTOR signaling). | 2 years
  Evaluate tissue collected at progression for activation state of signaling pathways that are known markers for endocrine resistance
Determine frequency when "multi-omic" profiling: proteomic and genomic profiling analysis of patient's tumor yields a target against which there is an FDA-approved agent or therapeutic regimen. | 2 years
  Evaluate frequency with which multiomic profiling analysis of patient's tumor identifies a target that can be treated by an FDA-approved agent or regimen
Determine percent of time multiomic profiling based treatment recommendation is different than treatment selected by the patient's physician once a patient shows progression after first line treatment with palbociclib or ribociclib | 2 years
  Evaluate percentage of time when treatment recommendations found with multiomic profiling is different than treatment selected by a patient's physician

OTHER OUTCOMES:
Perform RPPA based batch analysis of all samples at the end of this study to measure 50-100 protein signaling targets. Protein activation will be correlated with clinical response. | 2 years
  The data from this exploratory analysis will help generate hypotheses for future studies.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UHealth/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Abramson Cancer Center Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No